CLINICAL TRIAL: NCT04996225
Title: Effect of Aerobics and Balancing Exercises on Anxiety and Dizziness in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merit University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A,B E COVID 19
Record Dates: First submitted 2021-08-06; First posted 2021-08-09 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Corona Virus Infection
Keywords: Aerobics - Balance exercises -anxiety - dizziness disorder
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Finally, it could be concluded that aerobic exercise and balancing exercise with relaxation exercises decrease anxiety and dizziness in patients with COVID-19. So, it considered as effective, safe, cheap and successful adjunct treatment methods in reducing anxiety and dizziness in patients with COVID-19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A): (study group) (Experimental): Group (A): (study group) 15 patients received aerobics exercises and balancing exercises in addition to relaxation exercises for 4 weeks, 3sessions/week.
  Interventions: Other: Aerobics exercises, Balance exercises
- Group (B): (Control group) (Placebo Comparator): 2-Group (B): (Control group) 15 patients received relaxation exercises in the form of physical relaxation exercise for 4 weeks, 3 sessions/week. the participants who received aerobics exercises and balancing exercises in addition to relaxation exercises (experimental group A), showed significant decrease in anxiety and dizziness more than (placebo group B)
  Interventions: Other: Aerobics exercises, Balance exercises

INTERVENTIONS:
Other: Aerobics exercises, Balance exercises — Aerobic exercise, or endurance exercise, is a subdivision of physical exercise that improves cardiovascular and respiratory health. Additionally, it is generally assumed to increase well-being and reduce negative mood states such as anxiety and depression.

SUMMARY:
The recently emerged coronavirus named Severe Acute Respiratory Syndrome Coronavirus 2 (SARSCoV-2) is the newest threat to human health. It has already infected more than half a million people worldwide, leading to a lot of deaths. Patients with Coronavirus Disease 2019(COVID-19) will experience high levels of anxiety and low sleep quality due to isolation treatment. Purposes: Was to investigate the effect of aerobics and balancing exercises on anxiety and dizziness in patients with COVID-19. Subjects: Thirty anxiety and dizziness patients with COVID-19 aged from 45-65 years of both sexes, randomly divided into two groups, selected from outpatient clinic ,General

DETAILED DESCRIPTION:
In December 2019, a series of pneumonia cases of unknown cause emerged in Wuhan, Hubei, China, with clinical presentations greatly resembling viral pneumonia. Deep sequencing analysis from lower respiratory tract samples indicated a novel coronavirus, which was named 2019 novel coronavirus Disease (COVID-19). On February 12, 2020, WHO officially named the disease caused by the novel coronavirus as Coronavirus Disease 2019 (COVID-19),and by March 11th, 2020 when the number of countries involved was 114, with more than 118,000 cases and over 4000 deaths, the WHO declared the pandemic status

ELIGIBILITY:
Inclusion Criteria:

* Thirty patients with COVID-19
* Age between 45 -65 years
* Cooperative patient.
* All patients were referred from physician with the diagnosis of COVID-19

Exclusion Criteria:

* Overweigh patients with body mass index more than 30.
* Pregnant women.
* Cancer patients.
* Smokers
* Patients with chronic heart disease

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
SPSS for Windows, version 22 (SPSS Inc., Chicago, Illinois, USA) | one month
  Statistical analysis was carried out using SPSS for Windows, version 22 (SPSS Inc., Chicago, Illinois, USA). The P value is the degree of significant. A P value less than or equal to 0.05 was considered to be significant. Comparison between the mean values of different parameters in the two groups was performed using an unpaired t test. Comparison between pretreatment and post-treatment data in the same group was performed using a paired t test.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Essa, PHD, Study Chair — Lecturer of Biomechanics, Faculty of Physical Therapy, Deraya University, Minia,
Locations (1):
- Ahmed.Assem, Sohag, Egypt

REFERENCES:
- [Background] Lu H, Stratton CW, Tang YW. Outbreak of pneumonia of unknown etiology in Wuhan, China: The mystery and the miracle. J Med Virol. 2020 Apr;92(4):401-402. doi: 10.1002/jmv.25678. Epub 2020 Feb 12. No abstract available. PMID 31950516
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Rajeswari S, SanjeevaReddy N. Efficacy of Progressive Muscle Relaxation on Pregnancy Outcome among Anxious Indian Primi Mothers. Iran J Nurs Midwifery Res. 2019 Dec 27;25(1):23-30. doi: 10.4103/ijnmr.IJNMR_207_18. eCollection 2020 Jan-Feb. PMID 31956594
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Background] Chekroud SR, Gueorguieva R, Zheutlin AB, Paulus M, Krumholz HM, Krystal JH, Chekroud AM. Association between physical exercise and mental health in 1.2 million individuals in the USA between 2011 and 2015: a cross-sectional study. Lancet Psychiatry. 2018 Sep;5(9):739-746. doi: 10.1016/S2215-0366(18)30227-X. Epub 2018 Aug 8. PMID 30099000